CLINICAL TRIAL: NCT05729854
Title: The Effect of Acupressure on Shoulder Pain and Breastfeeding Self-efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Kubra Turkben, research assistant, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aiçu-ebe-KT-01
Record Dates: First submitted 2023-01-30; First posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Shoulder Pain
Keywords: cesarean; shoulder pain; acupressure; breast-feeding; Midwifery
MeSH Terms: conditions — Shoulder Pain; Breast Feeding | interventions — Acupressure; Complementary Therapies

STUDY DESIGN:
Intervention Model Description: experimental and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure group (Experimental): Acupressure will be performed by the researchers of the main, hand and body parts of the women in the experimental units.In the clinic where the study will be conducted, acupressure application hours were determined considering the analgesic treatment protocol applied. Acupressure will be applied at the 18th and 24th hours postpartum.
  Interventions: Other: acupressure ( traditional and complementary medicine)
- control group (No Intervention): Acupressure will not be applied to the control group. routine midwifery care.

INTERVENTIONS:
Other: acupressure ( traditional and complementary medicine) — Acupressure will be applied to the shoulders, hands and legs of the women in the experimental group by the researcher.
  Arms: acupressure group

SUMMARY:
In this study, for the first time in our country, acupressure will be examined on post-cesarean shoulder pain and breastfeeding self-efficacy by using a combination of shoulder (GB21), hand (LI4) and leg (ST36) points and applying acupressure as repeated sessions.

DETAILED DESCRIPTION:
After a cesarean delivery, pain causes patient dissatisfaction, impaired recovery, longer hospital stays, and delayed return to normal activities. The incidence of pain in the shoulder is high after surgery on the abdomen and its organs (visceral surgery). It has an incidence of 97% in thoracotomy, 71.4% in laparoscopy, and 40% in women who underwent cesarean section. Many studies in the review of shoulder pain after surgical procedures for the abdomen and its organs blame the phrenic nerve for transmission of shoulder pain and consider it a referred pain. Effective management of pain after childbirth will enable a woman to focus on early maternal duties and reduce the risk of persistent pain and depression.7 Pain interferes with babysitting and other activities of daily living. Therefore, postpartum pain management is critical to successful breastfeeding. Limited mobility after cesarean section may prevent the baby from taking an adequate position at the breast, and pain may inhibit the let-down reflex. Non-pharmacological treatments are useful because they are simple, effective and economical, reduce opioid consumption and increase patient satisfaction. Acupressure is a hand-mediated energy healing technique. Acupressure as a whole is a manually operated, needle-free, non-invasive, cost-effective and non-pharmacological healing intervention to improve patients' well-being. While the emergence of positive situations such as excitement or satisfaction increases breastfeeding self-efficacy; Negative states such as pain, fatigue, anxiety or stress reduce the perception of breastfeeding self-efficacy. Since the mother is in both the postpartum and postoperative period after the cesarean section, pain management is provided in the safest way for the mother and the baby; Supporting pharmacological treatment with non-pharmacological applications has an important place in midwifery care. This study is unique in that it is the first time in our country to examine acupressure on shoulder pain and breastfeeding self-efficacy after cesarean section by using a combination of shoulder (GB21), hand (LI4) and leg (ST36) points and applying acupressure as repeated sessions.

ELIGIBILITY:
Inclusion Criteria

* Those whose pain intensity is 45 mm or more according to the Vision Analogue Scale (VAS),
* Those who are disturbing and above according to the verbal category scale (SCS),
* Cesarean delivery by applying spinal anesthesia,
* who has an outdated, single and healthy newborn,
* 37-40 weeks of gestation,
* Between 18 and 45 years old,
* No fractures or dislocations in the shoulder,
* The absence of chronic pain in the shoulder,
* No history of trauma on the shoulder,
* No systemic and chronic diseases,
* No communication problems
* Women who agree to participate in the study will be sampled.

Exclusion Criteria:

* Cesarean delivery with general anesthesia
* Shoulder pain before cesarean section,
* Those who develop any complications related to the mother and the baby in the postpartum period (bleeding, hypertension, babies taken to the neonatal intensive care unit, etc.),
* Have a body mass index above 25 kg/m2,
* Have previous acupressure experience,
* Patients who consume caffeine (tea, coffee, chocolate...),
* If necessary, patients who underwent analgesia will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — patient having a cesarean section
Enrollment: 90 (Estimated)
Dates: Start 2023-02-20 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Visual Comparison Scale (Visual Analog Scale (VAS)) | one day
  In the evaluation of VAS, 0 mm = no pain, 100 mm refers to unbearable pain. On the scale, 0-44 mm shows mild pain, 45-74 mm shows moderate pain, and 75-100 mm shows severe pain

SECONDARY OUTCOMES:
Verbal Category Scale (SCS) | one day
  To describe the severity of pain on the scale, there are the words (1) mild, (2) disturbing, (3) severe, (4) very severe, (5) unbearable.
BREASTFEEDING SELF-EFFICACY SCALE SHORT FORM | one day
  The minimum score that can be obtained from the scale is 14, the maximum score is 70, and the scale has no breakpoint. An increase in the scale score means that breastfeeding self-efficacy is high.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Türkben, Principal Investigator — kturkben@agri.edu.tr

IPD SHARING:
Plan to Share IPD: No